CLINICAL TRIAL: NCT02058173
Title: "Pharmacoepidemiological Evaluation of Autophagy Inhibition in Treatment of HCV Patients Resistant to Standard Therapy. Pilot Study"
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Payam Peymani, PhD Student of pharmacoepidemiology,health policy reseach center,Shiraz University of Medical Sciences, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HP7-92; HP7-92 (Registry Identifier: HP7-92)
Record Dates: First submitted 2014-02-05; First posted 2014-02-07 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Hepatitis C Virus
MeSH Terms: conditions — Hepatitis C | interventions — Chloroquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- chloroquine (Experimental): 150 mg chloroquine and lacebo , one tablet daily for 2 month
  Interventions: Drug: 150 mg/daily chloroquine compare to placebo for 12 week; Drug: Chloroquine
- placebo (Experimental): 150 mg chloroquine and lacebo , one tablet daily for 2 month
  Interventions: Drug: 150 mg/daily chloroquine compare to placebo for 12 week; Drug: placebo

INTERVENTIONS:
Drug: 150 mg/daily chloroquine compare to placebo for 12 week
Drug: Chloroquine
  Arms: chloroquine
Drug: placebo
  Arms: placebo

SUMMARY:
The purpose of this study is to assess the efficacy of Chloroquine comparing with placebo for treatment of non- response HCV patients.. In this triple blind pilot study, 20 patients with confirmed chronic hepatitis C will be randomize into treatment group (Chloroquine 150 mg daily, for 8 weeks) or control group (placebo once daily, for 8 weeks). Patients who have receiving anti neoplastic, anti viral or Immunomedullator drugs during 6 months prior to study, have co-infection Hepatitis A,C,D or HIV, severe liver or renal dysfunction, are pregnant or breast fed, or refuse to sign informed consent will be excluded.. At the end of therapy (12 weeks) and at baseline, first, second and third month after receiving drug and placebo HCV Virus load, CBC LFT and biochemical parameters will be evaluated and compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* patients who failed to achieve a decline of 2 log HCV RNA IU/ml after 12 weeks of treatment
* who never achieved undetectable HCV RNA during treatment of a minimum duration of 24 weeks

Exclusion Criteria:

* Receiving anti neoplasm, anti viral or immunomedulator drugs during 6 months prior to study
* coinfection with Hepatitis A,C,D viruses or HIV
* Severe dysfunction of liver and kidney
* pregnancy
* breast feeding
* refusing to give informed consent
* active Alcohol user
* presence of decompensate cirrhosis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2014-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Loss of HCV RNA at end of treatment which is 8 weeks | march 2014

SECONDARY OUTCOMES:
Two log decrease in HCV RNA at the end of treatment | july 2014

OTHER OUTCOMES:
ALT response which is significant decrease in ALT-(biochemical response during Treatment) | july 2014

CONTACTS AND LOCATIONS:
Overall Officials: Kamran B Lankarani, M.D, Study Chair — Health policy research center
Locations (1):
- Health Policy Research Center, Shiraz, Fars, Iran